CLINICAL TRIAL: NCT06872489
Title: Expanded Access Protocol for the Use of SL-28 in the Treatment of Advanced Solid Tumors
Status: Available | Type: Expanded Access
Sponsor: Second Life Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: SL28-NBL-G4407
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma in Children; Neuroblastoma, Recurrent, Refractory; Advanced Cancer; Advanced Malignant Neoplasm; Prostate Cancer Patients With Bone Metastasis; Lung Cancer Non-Small Cell Cancer (NSCLC); Lung Cancer - Non Small Cell; Gastrointestinal Cancers; Head and Neck Cancer; Pancreatic Cancer
MeSH Terms: conditions — Neuroblastoma; Recurrence; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Pancreatic Neoplasms

INTERVENTIONS:
Biological: SL-28. — Allogeneic, non-HLA matched, Leucocyte-Tells-based therapy

SUMMARY:
This is an Expanded Access Program (EAP) that will give the participants access to the drug SL-28 before it is approved by the FDA. Participants in this study will have Advanced Solid Tumors who failed to respond to standard therapy (chemotherapy, immunotherapy) or developed progressive disease at any phase of standard therapy.

Researchers think the SL-28 will be effective because SL-28 has a direct activity against different types of tumors.

SL-28 is a cell-based therapy, based on leukocytes isolated from healthy donors and are activated through the proprietary process. After quality assessment (sterility, viable cell count, purity, and absence of infectious diseases), they are stored at -80°C until use. Upon need, the SL-28 is thawed, followed by checking their viability, count, and sterility. Adult and older adult patients aged 18 to 65+ who meet the eligibility criteria will be included in the study. Patients receive SL-28 IV once daily on days 1-5 and 8-12. Based on the patient's response, the need for additional injections will be evaluated. If improvements in the patient's condition are confirmed by MRI, further injections can continue on a rate 5 days a week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with locally advanced or metastatic solid tumor confirmed by histopathology;
* Having at least one evaluable or measurable lesion according to the solid tumor response Evaluation Criteria (RECIST 1.1);
* For patients with relapsed/refractory neuroblastoma with original diagnosis based on tumor histopathology, Karnofsky or Lansky performance status of ≥ 50%;
* ECOG Performance Status from 0 or 3;
* The expected survival time is more than 12 weeks;
* 2 to 65+ old, gender is not limited;
* The subjects gave informed consent to the study before participating in, and voluntarily signed informed consent;
* Be able to comply with trial and follow-up procedures;
* Adequate bone marrow and organ function;
* Patients who have progressed, recurrent or refractory disease after first-line treatment (failure to obtain complete or partial remission after recent treatment);
* Fertile women must agree to abstain from sex (abstaining from heterosexual intercourse)or use a highly effective method of contraception for at least one week from the time they sign an informed consent form until the last dose of the study drug.
* The blood HCG test must be negative within 7 days before the start of the study treatment, and must be non-lactating;
* For male patients whose partner is a woman of reproductive age, they must agree to abstain from sex for at least one week from signing the informed consent until the last dose of the study drug, or to use a highly effective method of contraception.
* Immunotherapy: At least 42 days after completing any type of immunotherapy, including immune checkpoint;
* Radiation therapy: 60 days should have elapsed in the case of completing radiation.
* Cytokine therapy (e.g. G-CSF, GM-CSF, IL-6, IL-2): must be discontinued a minimum of 7 days prior to SL-28 therapy.

Exclusion Criteria:

* Untreated or active primary central nervous system (CNS) tumor or metastasis;
* Patients diagnosed of having primary and secondary immunodeficiencies;
* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Arterial/venous thrombosis events that occurred in the 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Known allergy to any of the agents or their ingredients used in this study;
* Patients who are on hemodialysis;
* Pregnant or breast-feeding women; fertility patients who are unwilling or unable to take effective contraceptive measures;
* Patients with untreated positive blood cultures or progressive infections.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult